CLINICAL TRIAL: NCT04964856
Title: Enhanced Recovery After Surgery Exercise Improve Perioperative Frailty of Patients Undergoing Elective Surgery:a Randomized Controlled Clinical Trial
Brief Title: Enhanced Recovery After Surgery Exercise Improve Perioperative Frailty
Acronym: EEIPF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, Director of Department of Anesthesiology, The First Affiliated Hospital of Chongqing Medical University, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYYYMZK-E
Record Dates: First submitted 2021-03-19; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: ERAS; Frailty
Keywords: ERAS; Frailty; Exercise; Activity
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS exercise in perioperative period. (Experimental): The patients take ERAS exercise from hospitalization to 30 days after operation.
  Interventions: Behavioral: ERAS exercise
- No ERAS exercise in perioperative period. (Sham Comparator): The patients do not take ERAS exercise in perioperative period.
  Interventions: Behavioral: No ERAS exercise

INTERVENTIONS:
Behavioral: ERAS exercise — Take ERAS exercise twice a day from hospitalization to 30 days after surgery
  Arms: ERAS exercise in perioperative period.
Behavioral: No ERAS exercise — Don't take ERAS exercise in perioperative period
  Arms: No ERAS exercise in perioperative period.

SUMMARY:
A randomized, controlled, clinical trial on the efficacy of ERAS exercise improve perioperative frailty in patients undergoing elective laparoscopic colorectal surgery

Objective to evaluate the efficacy of ERAS exercise improve perioperative frailty in patients undergoing elective laparoscopic colorectal surgery

Participants: Patients undergoing elective laparoscopic colorectal surgery over 18 years old.

The research intervention was ERAS exercise

The study design was a randomized, parallel controlled trial

ERAS exercise in perioperative period as the experimental group. No ERAS exercise group was the control group.

The sample size was estimated according to the main efficacy index ( the attenuation of frailty after 7 days surgery) of this study. It was assumed that the attenuation of frailty in the ERAS exercise group was better than that of the control group. The parameters were set as test level (alpha) of 0.050 using a two-sided two-sample unequal-variance t-test, β = 0.9, according to the results of previous clinical trials and combined with literature, the population mean difference was 0.6 with standard deviations of 0.8 for the experimental group and 0.8 for the control group. the experimental group: the control group was 1:1, 39 cases in each group, considering the 20% shedding rate, 49 cases in the experimental group and 49 cases in the control group were selected.

1. The experimental group The patients take ERAS exercise from hospitalization to 30 days after operation.
2. The control group The patients do not take ERAS exercise in perioperative period.

Efficacy evaluation

1. The primary endpoint of the study was the attenuation of frailty via Frailty Phenotype (FP) between before surgery and 7days, 30 days after surgery.
2. Secondary endpoints included the 6-minute walk test (6MWT),nutritional risk screening (NRS2002), anxious and depressive states, activities of daily living (ADL),postoperative complications and mortality,short-term recovery quality,postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving elective laparoscopic colorectal surgery.
* 18≤age≤100 years old, no gender limit;
* The ASA score is between I and Ⅲ;
* Clearly understand and voluntarily participate in the study, and sign an informed consent form.

Exclusion Criteria:

* Emergency surgery;
* Those with a history of cognitive dysfunction;
* Those with a history of neuromuscular diseases,;
* American Society of Anesthesiologists class ⩾IV;
* Those with a history of spontaneous pneumothorax, coagulation dysfunction,
* Acute and systemic infectious diseases, moderate or higher fever;
* Pregnant women;
* History of drug abuse;
* Those who judged by the physician in charge to be unsuitable for ERAS-exercise;
* Other severe cardio-pulmonary diseases that would affect the 6MWD
* Those failure to obtain informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Frailty status | Change from Baseline Fried's Frailty Phenotype scores at 30 days postoperatively
  Frailty status (i.e. robust, prefrail or frail) measured using the Fried's Frailty Phenotype (FP) scores. Frailty scores from 0 to 5 (i.e., 1 point for each component; 0 = best to 5 = worst) and represent robust (0), pre-frail (1-2), and frail (3-5) health status.

SECONDARY OUTCOMES:
Change in gait speed | baseline, at 30 days postoperatively
  This outcome will be measured using the 5-meter walk test.
Handgrip strength | baseline, at 30 days postoperatively
  Handgrip strength will be measured using a dynamometer.
Perioperative functional capacity | baseline, at 30 days postoperatively
  The 6-minute walk distance (6MWD) test is a non-encouraged test performed in a 30 meters long flat corridor, where the participant is instructed to walk as far as possible, back and forth around two cones, with the permission to slow down, rest, or stop if needed. Ambulation was assessed via the 6MWD test following standardized procedures by measuring the 6MWD in meters. Participants were not permitted to use assistive devices (walker, long leg braces, or short leg braces) during the 6MWD test. Participants with confirmed loss of ambulation at a particular visit were assigned a 6MWD result of 0.
Patient mood state | baseline and 7th day postoperatively
  This outcome will be assessed using Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.
Nutritional status | baseline, at 30 days postoperatively
  This outcome will be assessed using Nutritional Risk Screening 2002 (NRS-2002): The patients were classified as being nutritionally risk (NRS+): total score ≥ 3 or nutritionally risk-free (NRS-): total score < 3 according to NRS 2002 results.
Short-term recovery quality | baseline, 1st, 2nd, 3rd and 7th day postoperatively
  This outcome will be measured using 9-item quality of recovery(QoR-9) score.The QoR-9 is a 9-item score evaluating both physical and mental well-being by assessing five dimensions: emotional state, physical comfort, psychological support, physical independence and pain. Each of the 9 items are scored by the patient from 0 (worst score) to 2 (best score), giving a lowest possible score of 0 (worst outcome), and a highest possible score of 18 (best outcome).
Postoperative Complications | 30 days postoperatively
  Postoperative Complications evaluated by Clavien- Dindo Score.Nine domains are evaluated: Pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, wound, haematological and pain. Each domain is graded between grade I and V (death of a patient).
Postoperative 30-day mortality | 30 days postoperatively
  Rate of Mortality among study patients
Highest VAS Pain Score at Rest | baseline, 1st, 2nd, 3rd and 7th day postoperatively
  Post-operative pain scores at rest, as assessed by Visual Analog Pain Scale (VAS) will be the primary outcome measured. Postoperative pain at rest will be defined as the highest VAS pain score reported by each patient at any time. Pain score is from 0 (no hurt) to 10 (hurts worst).
Highest VAS Pain Score during Exercise | baseline, 1st, 2nd, 3rd and 7th day postoperatively
  Post-operative pain scores during Exercise, as assessed by Visual Analog Pain Scale (VAS) will be the primary outcome measured. Postoperative pain during Exerciset will be defined as the highest VAS pain score reported by each patient at any time. Pain score is from 0 (no hurt) to 10 (hurts worst).

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Yang F, Yuan Y, Liu W, Tang C, He F, Chen D, Xiong J, Huang G, Qian K. Effect of prehabilitation exercises on postoperative frailty in patients undergoing laparoscopic colorectal cancer surgery. Front Oncol. 2024 Sep 12;14:1411353. doi: 10.3389/fonc.2024.1411353. eCollection 2024. PMID 39328202